CLINICAL TRIAL: NCT02508597
Title: Brief Tobacco Cessation Counselling: Mini Train-the-trainers Program Among Physicians in Guangdong, China
Brief Title: Brief Tobacco Cessation Counselling: Mini Train-the-trainers Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Chair Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MiniTTT
Record Dates: First submitted 2015-07-08; First posted 2015-07-27 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Smoking
Keywords: Smoking cessation intervention
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physicians receiving smoking cessation training (Other): On the training day, the investigators will explain at the beginning of the workshop the purpose of the training, and the details of the brief smoking cessation intervention to all physicians who attend the training workshop.
  Interventions: Other: Physicians receiving smoking cessation training

INTERVENTIONS:
Other: Physicians receiving smoking cessation training — On the training day, the investigators will explain at the beginning of the workshop the purpose of the training, and the details of the brief smoking cessation intervention to all physicians who attend the training workshop.

SUMMARY:
Physicians play a critical role in reducing tobacco use by advising smoking patients to quit. After receiving such advice to quit smoking, patients were more likely to report trying to quit, quitting for at least 24 hours, making more quit attempts, and having more successful quitting outcomes compared with those who received no such advice. On the other hand, most physicians are not performing smoking cessation counselling, and miss the opportunities to advise patients to quit smoking. One of the common reasons is the lack of time. Physicians are busy and cannot afford even one minute to advice their patients to quit smoking. Other barriers include lack of training and experience, lack of knowledge and skills, no awareness about the benefits and effects of physicians' advice, no incentives and no support or requirement from hospital management that they have to do it.

We designed a brief smoking cessation counselling model (AWARD) which takes only 10-20 seconds. We will train the physicians to perform the AWARD cessation counselling model in clinic, and encourage them to participate in our brief smoking cessation intervention project using the randomized controlled trail (RCT) design and to train more peer physicians to perform brief smoking cessation counseling. We propose to investigate the effect of the training program on physicians' knowledge of tobacco cessation, practice of performing cessation counselling, and attitudes toward tobacco control policies.

DETAILED DESCRIPTION:
Participating hospitals/clinics will invite 100-120 internal medicine physicians to take part in the brief smoking counselling intervention project and participate in a half-day mini TTT training program. The training will cover the following topics:

* Goal and the details of the brief smoking counselling intervention;
* Objective of the mini TTT training program;
* Tobacco epidemic and control measures in China and the world;
* Physicians' role in tobacco control;
* Health risks of smoking, secondhand smoke exposure;
* WHO FCTC (Framework Convention on Tobacco Control) and the MPOWER measures;
* Brief smoking cessation counselling (AWARD model), and counselling skill with practice;
* Placebo counselling and counselling skill with practice.

On the training day, the investigators will explain at the beginning of the workshop the purpose of the training, and the details of the brief smoking cessation intervention to all physicians who attend the training workshop. The investigators will explain that the participation is totally voluntary, and the participants will be invited to complete a paper-and-pencil survey before and right after the training workshop, perform smoking cessation counselling or placebo counselling among patients at their clinics, and complete online survey at 6- and 12-month follow-up. Agreement to participate in the training program will be considered as consent and participants are required to sign a written consent form.

At the end of the workshop, participants should be confident to perform brief smoking cessation counselling and placebo counselling for patients.

We hypothesize that the training program will increase the participants' knowledge level of smoking and secondhand smoke exposure and the important role of physicians in tobacco control, increase their skill and confidence of performing smoking cessation counselling, and generate stronger support for tobacco control policies.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine physicians from participating hospitals/clinics.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
KAP change from baseline at 6-month follow-up | 6-month follow-up
  Use questionnaire to measure the change of "Knowledge of smoking, secondhand smoke exposure, and the role of physicians in tobacco control", "Attitudes toward tobacco control policies" and "Practice of smoking cessation counseling" (KAP)
KAP change from baseline at 12-month follow-up | 12-month follow-up
  Use questionnaire to measure the change of "Knowledge of smoking, secondhand smoke exposure, and the role of physicians in tobacco control", "Attitudes toward tobacco control policies" and "Practice of smoking cessation counseling" (KAP)

SECONDARY OUTCOMES:
Satisfaction of the mini TTT workshop | 24 months
  A questionnaire will be completed by workshop participants to measure satisfaction of mini TTT workshop after each workshop
Number of peer physicians the participants trained | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- 5/F William MW Mong Block, LKS Faculty of Medicine Building, 21 Sassoon Road, Pokfulam, Hong Kong, Guangdong, China